CLINICAL TRIAL: NCT03808623
Title: Non-interventional Study to Evaluate the Safety and Performance of NOVOCART® Basic and the Clinical Outcome of MAC With NOVOCART® Basic in Patients Treated for Cartilage Defects in the Knee.
Brief Title: Non-interventional Study With NOVOCART® Basic in Patients Treated for Cartilage Defects in the Knee With MAC
Acronym: NBasic
Status: Completed | Type: Observational
Sponsor: Tetec AG (Industry)
Collaborators: Aesculap AG (Industry); Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1712
Record Dates: First submitted 2019-01-08; First posted 2019-01-17 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Cartilage Diseases
Keywords: cartilage defect; knee; MAC (Matrix associated chondrogenesis)
MeSH Terms: conditions — Cartilage Diseases; Mycobacterium avium-intracellulare Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MAC with NOVOCART Basic — NOVOCART® Basic is a biphasic, collagen-based matrix to support the biological reconstruction of localized and full-thickness cartilage damages after treatment with bone marrow stimulation techniques (microfracture). The procedure is called matrix associated chondrogenesis (MAC). It is a single-step procedure.
  NOVOCART® Basic is tailored to fit the prepared defect size and is inserted in the defect area after microfracture. The NOVOCART® Basic device component is fully resorbed over a period of a few months as new reparative cartilage tissue is generated and integrated with the surrounding host tissue.
  Other Names: MAC

SUMMARY:
Retrospective, multicenter, single arm, non-interventional study to assess the safety and Performance of NOVOCART Basic and the clinical outcome of MAC with NOVOCART Basic in patients treated for cartilage defects in the knee.

DETAILED DESCRIPTION:
This study is a multi-center, single arm, non-interventional study to assess the safety and performance of NOVOCART® Basic and the clinical outcome of MAC with NOVOCART® Basic in patients treated for cartilage defects in the knee. In this study data will be collected retrospectively from patient files of adult and pediatric patients who had received an MAC with NOVOCART® Basic for cartilage defects in the knee according to medical practice. In addition, at the time when a patient consents to participate in the study, he/she will have to fill-out questionnaires on current symptoms and knee function, quality of life, satisfaction with treatment and subsequent surgical interventions on the target knee performed outside the study site, i.e. the duration of follow-up is not standardized. All clinical sites having treated more than 8 patients with NOVOCART® Basic between 2014 and 2017 will be contacted for participation. Participating clinical sites will be asked to collect informed consent from their patients to document relevant data from their medical charts and to complete the questionnaires. Consenting patients will send the signed informed consent form(s) and the completed questionnaires back to the study site. The date of questionnaire completion is regarded the end of observation for an individual patient. For data documentation, a medical documentation specialist authorized by TETEC AG will be given access to the patient files, the informed consent forms, and the completed questionnaires. The relevant data will be entered directly into an electronic database by the medical documentation specialist. Only data from patients who have given informed consent to study participation will be documented. If available, post-MAC MRIs will be collected and reviewed by independent experts.

ELIGIBILITY:
Inclusion Criteria:

* for the biological reconstruction of localized full-layer cartilage damage (III and IV degree defects pursuant to the ICRS classification) in the knee joint.
* Treatable defects include:
* Cartilage damage caused by trauma
* Defects due to osteochondrosis dissecans
* Smaller focally-limited, degenerative cartilage damage
* Patients aged between 18 and 55 years
* Cartilage defect sizes from 1.5 to 4 cm²
* Deep osseous substance defects require prior osseous reconstruction. The indication should be confirmed using arthroscopy.

Exclusion Criteria:

* Patients with known allergies to bovine collagen.
* Infected joints or infected wounds/areas near the joint, arthritis or inflammatory joint diseases of any type are contraindicated.
* More than two corresponding cartilage defects
* Instability of the knee, subtotal/total meniscus resection
* Varus/valgus malpositions (corrective surgery required in such cases)
* Haemorrhagic diathesis of various origins
* Applications which are not listed in the Indications section.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: All patients (adult and pediatric) who have received an MAC with NOVOCART® Basic in the knee are eligible for this study, provided that they have given their informed consent for data collection and the involved clinical site has agreed to participate.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety of NOVOCART® Basic | Up to 5 years
  Number of participants with treatment related adverse device effects or adverse events related to the procedure involved

SECONDARY OUTCOMES:
Rate of therapy change | Up to 5 years
  Rate of therapy change (other surgical cartilage repair modality applied to the MAC treated defect(s))
Rate of adverse device effects | Up to 5 years
  Number of treatment related adverse device effects
Rate of device deficiencies | Up to 5 years
  Number of device deficiencies
Rate of adverse events related to the procedure involved | Up to 5 years
  Number of adverse events related to the procedure involved
KOOS | Up to 5 years
  Questionnaire: Knee injury and Osteoarthrisits Outcome Score (KOOS)(KOOS5 and subscores)
IKDC | Up to 5 years
  Questionnaire: International Knee Documentation Committee (IKDC2000) subjective score
EQ-5D-5L | Up to 5 years
  Quality of life (EQ-5D-5L index)
Patient satisfaction with treatment | Up to 5 years
  5 questions to patient satisfaction with treatment
MRI if available | Up to 5 years
  Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score will be used for assessment of the in vivo performance, if post-MAC MRIs are available from clinical routine

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Waibl, MD, Principal Investigator — Cartilage Care
Locations (3):
- Theresienkrankenhaus und St. Hedwig-Klinik GmbH, Mannheim, Baden-Wurttemberg, Germany
- Switzerland (2):
  - Praxisklinik Rennbahn AG, Muttenz, Cantone of Basel-Landschaft
  - Cartilage Care, Bern, Cantone of Bern